CLINICAL TRIAL: NCT05431075
Title: Bismuth-containing Quadruple Therapy for Helicobacter Pylori First-line Treatment: A Multicenter Randomized Clinical Trial of Different Tetracycline Doses and Frequencies.
Brief Title: Bismuth-containing Quadruple Therapy for Helicobacter Pylori First-line Treatment of Different Tetracycline Doses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Peking University Care Luzhong Hospital (Other); Yuncheng Traditional Chinese Medicine Hospital (Other); Taierzhuang District People's Hospital (Other); Zhengzhou Central Hospital (Other); Zibo Central Hospital (Other Government)
Responsible Party: Principal Investigator, Xiuli Zuo, Director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SDU-QILU-G004
Record Dates: First submitted 2022-06-18; First posted 2022-06-24 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; tetracycline; Bismuth-containing quadruple regimen
MeSH Terms: interventions — Amoxicillin; Esomeprazole

STUDY DESIGN:
Intervention Model Description: This trial is a multi-center, open-label, non-inferiority, randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tid group (Experimental): Tid group: Amoxicillin 1000mg bid+ Tetracycline 500mg tid+ Bismuth + Esomeprazole 20mg bid
  Interventions: Drug: Amoxicillin; Drug: Tetracycline tid; Drug: Bismuth Potassium Citrate; Drug: Colloidal Bismuth Pectin; Drug: Esomeprazole 20mg
- Qid group (Active Comparator): Qid group: Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth + Esomeprazole 20mg bid
  Interventions: Drug: Amoxicillin; Drug: Tetracycline qid; Drug: Bismuth Potassium Citrate; Drug: Colloidal Bismuth Pectin; Drug: Esomeprazole 20mg

INTERVENTIONS:
Drug: Amoxicillin — Included in quadruple eradication medication.
Drug: Tetracycline tid — Included in quadruple eradication medication.
  Arms: Tid group
Drug: Tetracycline qid — Included in quadruple eradication medication.
  Arms: Qid group
Drug: Bismuth Potassium Citrate — Included in quadruple eradication medication.
Drug: Colloidal Bismuth Pectin — Included in quadruple eradication medication.
Drug: Esomeprazole 20mg — Included in quadruple eradication medication.

SUMMARY:
The researchers collect treatment-naive H.pylori-positive patients from the outpatient clinic. The subjects were randomized to receive a dose and frequency of tetracycline 500mg tid or qid of bismuth quadruple eradication therapy. 6-8 weeks after treatment, the subjects will re-take the 13C-urea breath test. Calculate the eradication rates, adverse reaction rates, patient compliance and cost-effectiveness index of each group.

DETAILED DESCRIPTION:
The researchers collect treatment-naive H.pylori-positive patients from the outpatient clinic. If the subject meets the selection criteria but not the exclusion criteria, and signs an informed consent form, the researchers randomized the subjects in groups: subjects received a dose and frequency of tetracycline 500mg tid or qid of bismuth-containing quadruple eradication therapy. The medication of groups are as follows. 6-8 weeks after the eradication treatment, the subjects will review the 13C-urea breath test, and the researcher records the results.

After all subjects were tested, the eradication rates, adverse reaction rates, patient compliance and cost-effectiveness index of each group were calculated.

According to the course of treatment, it is randomized into a tid treatment group and a qid treatment group. The two groups of bismuth quadruple regimens are the same, as follows:

Tid group: Amoxicillin 1000mg bid+ Tetracycline 500mg tid+ Bismuth + Esomeprazole 20mg bid Qid group: Amoxicillin 1000mg bid+ Tetracycline 500mg qid+ Bismuth + Esomeprazole 20mg bid

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70.
* Patients with H.pylori infection (Positive for rapid urease test or 13C/14C-urea breath test).
* Patients who have never received H. pylori eradication treatment.

Exclusion Criteria:

* Patients with serious underlying diseases, such as liver insufficiency (Aspartate aminotransferase or alanine aminotransferase greater than 1.5 times the normal value), renal insufficiency (Cr≥2.0mg/dL or glomerular filtration rate <50 ml/min), immunosuppression, malignant tumors, Coronary heart disease or coronary artery stenosis ≥75%.
* Patients who are pregnant or lactating or unwilling to take contraceptive measures during the trial.
* Patients with active gastrointestinal bleeding.
* Patients with a history of upper gastrointestinal surgery.
* Patients allergic to treatment drugs.
* Patients with medication history of bismuth agents, antibiotics, proton pump inhibitor and other drugs within 4 weeks
* Patients with other behaviors that may increase the risk of illness, such as alcohol and drug abuse
* Patients who are unwilling or incapable to provide informed consents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Eradication rate | Immediately after follow-up check.
  Both intention to treat (ITT) and per-protocol (PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in two groups. The ITT analysis includes all randomly assigned patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
Rate of adverse reactions | Immediately after follow-up check.
  Rate of adverse reactions
Patient compliance | Immediately after follow-up check.
  Good compliance is defined as the actual dosage is within the range of 80%-100% of the dosage that should be taken.
Cost-effectiveness index | Immediately after follow-up check.
  Ratio of costs to effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (6):
- China (6):
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Qilu hosipital, Jinan, Shandong
  - Taierzhuang District People's Hospital, Taierzhuang, Shandong
  - Yuncheng Hospital of Traditional Chinese Medicine, Yuncheng, Shandong
  - PKUCare Luzhong Hospital, Zibo, Shandong
  - Zibo Central Hospital, Zibo, Shandong

REFERENCES:
- [Background] Hooi JKY, Lai WY, Ng WK, Suen MMY, Underwood FE, Tanyingoh D, Malfertheiner P, Graham DY, Wong VWS, Wu JCY, Chan FKL, Sung JJY, Kaplan GG, Ng SC. Global Prevalence of Helicobacter pylori Infection: Systematic Review and Meta-Analysis. Gastroenterology. 2017 Aug;153(2):420-429. doi: 10.1053/j.gastro.2017.04.022. Epub 2017 Apr 27. PMID 28456631
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Gisbert JP, Kuipers EJ, Axon AT, Bazzoli F, Gasbarrini A, Atherton J, Graham DY, Hunt R, Moayyedi P, Rokkas T, Rugge M, Selgrad M, Suerbaum S, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study Group and Consensus panel. Management of Helicobacter pylori infection-the Maastricht V/Florence Consensus Report. Gut. 2017 Jan;66(1):6-30. doi: 10.1136/gutjnl-2016-312288. Epub 2016 Oct 5. PMID 27707777
- [Background] Ding SZ, Du YQ, Lu H, Wang WH, Cheng H, Chen SY, Chen MH, Chen WC, Chen Y, Fang JY, Gao HJ, Guo MZ, Han Y, Hou XH, Hu FL, Jiang B, Jiang HX, Lan CH, Li JN, Li Y, Li YQ, Liu J, Li YM, Lyu B, Lu YY, Miao YL, Nie YZ, Qian JM, Sheng JQ, Tang CW, Wang F, Wang HH, Wang JB, Wang JT, Wang JP, Wang XH, Wu KC, Xia XZ, Xie WF, Xie Y, Xu JM, Yang CQ, Yang GB, Yuan Y, Zeng ZR, Zhang BY, Zhang GY, Zhang GX, Zhang JZ, Zhang ZY, Zheng PY, Zhu Y, Zuo XL, Zhou LY, Lyu NH, Yang YS, Li ZS; National Clinical Research Center for Digestive Diseases (Shanghai), Gastrointestinal Early Cancer Prevention & Treatment Alliance of China (GECA), Helicobacter pylori Study Group of Chinese Society of Gastroenterology, and Chinese Alliance for Helicobacter pylori Study. Chinese Consensus Report on Family-Based Helicobacter pylori Infection Control and Management (2021 Edition). Gut. 2022 Feb;71(2):238-253. doi: 10.1136/gutjnl-2021-325630. Epub 2021 Nov 26. PMID 34836916
- [Background] Lv ZF, Wang FC, Zheng HL, Wang B, Xie Y, Zhou XJ, Lv NH. Meta-analysis: is combination of tetracycline and amoxicillin suitable for Helicobacter pylori infection? World J Gastroenterol. 2015 Feb 28;21(8):2522-33. doi: 10.3748/wjg.v21.i8.2522. PMID 25741163
- [Background] Marko D, Calvet X, Ducons J, Guardiola J, Tito L, Bory F; GRESCA (Group for Eradication Studies from Catalonia and Aragon). Comparison of two management strategies for Helicobacter pylori treatment: clinical study and cost-effectiveness analysis. Helicobacter. 2005 Feb;10(1):22-32. doi: 10.1111/j.1523-5378.2005.00288.x. PMID 15691312
- [Background] Calvet X, Montserrat A, Guell M, Vergara M, Gene E. Ranitidine-bismuth citrate, tetracycline and metronidazole followed by triple therapy as alternative strategy for Helicobacter pylori treatment: a pilot study. Eur J Gastroenterol Hepatol. 2004 Oct;16(10):987-90. doi: 10.1097/00042737-200410000-00006. PMID 15371921
- [Background] Xie Y, Zhu Z, Wang J, Zhang L, Zhang Z, Lu H, Zeng Z, Chen S, Liu D, Lv N; the Chinese Study Group on Helicobacter pylori, Chinese Society of Gastroenterology. Ten-Day Quadruple Therapy Comprising Low-Dose Rabeprazole, Bismuth, Amoxicillin, and Tetracycline Is an Effective and Safe First-Line Treatment for Helicobacter pylori Infection in a Population with High Antibiotic Resistance: a Prospective, Multicenter, Randomized, Parallel-Controlled Clinical Trial in China. Antimicrob Agents Chemother. 2018 Aug 27;62(9):e00432-18. doi: 10.1128/AAC.00432-18. Print 2018 Sep. PMID 29914954
- [Background] Zhang J, Han C, Lu WQ, Wang N, Wu SR, Wang YX, Ma JP, Wang JH, Hao C, Yuan DH, Liu N, Shi YQ. A randomized, multicenter and noninferiority study of amoxicillin plus berberine vs tetracycline plus furazolidone in quadruple therapy for Helicobacter pylori rescue treatment. J Dig Dis. 2020 May;21(5):256-263. doi: 10.1111/1751-2980.12870. Epub 2020 Jun 9. PMID 32348007
- [Derived] Ding YM, Zhang QM, Li RL, Han ZX, Zhao Q, Xu LD, Wang KY, Nan XP, Duan M, Zeng SY, Kong QZ, Wang H, Wu XQ, Zhang N, Li YQ, Zuo XL, Li YY. Tetracycline Three Times Daily Versus Four Times Daily in Bismuth-Containing Quadruple Therapy as the First-Line Treatment of Helicobacter pylori Infection: A Multicenter, Noninferiority, Randomized Controlled Trial. Helicobacter. 2024 Jul-Aug;29(4):e13121. doi: 10.1111/hel.13121. PMID 39097924